CLINICAL TRIAL: NCT03984916
Title: Interventional Study for the Comparison of the Bioavailability of Three Hesperidin Extracts (HESPERIDIN).
Brief Title: Study of the Bioavailability of Three Hesperidin Extracts.
Acronym: HESPERIDIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technological Centre of Nutrition and Health, Spain (Other)
Collaborators: Fundació Eurecat (Other); Hospital Universitari Sant Joan de Reus (Other); University Rovira i Virgili (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: HESPERIDIN
Record Dates: First submitted 2019-06-07; First posted 2019-06-13 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Biological Availability
Keywords: hesperidin; orange extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The appearance of the interventions is identical, appearing in capsules of identical appearance and with a numerical code.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hesperidin Pharma (Active Comparator): 500 mg of sweet orange extract with a mixture of hesperidin isomers -S and -R. The approximate particle size is less than 100 µm for the 90% of the extract, and of 10 µm for 10% of the extract.
  Interventions: Dietary Supplement: Hesperidin Pharma
- Hesperidin Pharma_M (Active Comparator): 500 mg of sweet orange extract with a mixture of hesperidin isomers -S and -R. The size of 90% of particles is less than 10 µm.
  Interventions: Dietary Supplement: Hesperidin Pharma_M
- Cardiose (Experimental): 500 mg of sweet orange extract with more than 90% of the isomer -S. The size of the 90% of particles is less than 10 µm.
  Interventions: Dietary Supplement: Cardiose

INTERVENTIONS:
Dietary Supplement: Hesperidin Pharma — Two capsules with 250 mg of sweet orange extract with a mixture of hesperidin isomers -S and -R.
  Arms: Hesperidin Pharma
Dietary Supplement: Hesperidin Pharma_M — Two capsules with 250 mg of sweet orange extract each with a mixture of hesperidin isomers -S and -R and micronized.
  Arms: Hesperidin Pharma_M
Dietary Supplement: Cardiose — Two capsules with 250 mg of sweet orange extract each with more than 90% of hesperidin as isomer -S and micronized.
  Arms: Cardiose

SUMMARY:
The flavonoid hesperidin is present abundantly in citrus fruits and citrus juices. The results of numerous studies suggest that hesperidin perform several beneficial effects on health, including antitumor, antioxidant, anti-inflammatory, hypocholesterolemic and hypoglycemic effects as well as decreasing blood pressure.

There are two isomers of hesperidin, -S and -R, being the predominant form in nature the isomer -S. However, currently commercialized hesperidin consists of a mixture of both isomers due to the extraction process of the hesperidin from natural sources.

The presence of the rutin disaccharide conjugated to the hesperidin molecule is responsible that most of the ingested hesperidin is metabolized by bacteria in the colon through the enzymatic activity α-rhamnosidase, being this enzymatic activity the limiting step of the hydrolysis and absorption of hesperidin. It has been suggested that the low levels of this enzymatic activity in the gut microbiota is the cause of the low bioavailability of hesperidin and also, at least in part , of the high interindividual variability that exists in the absorption of this compound.

The micronization process in order to decrease the size of the hesperidin particles is presented as a way to increase the bioavailability of hesperidin. Another way to increase the absorption of hesperidin that is proposed in this study is to increase the proportion of the isomer -S in the extracts of hesperidin, since being the isomer that mostly occurs in nature, the gut microbiota will have a greater capacity of metabolism for this isomer.

On this basis the present hypothesis is posed: the administration of hesperidin formed mainly by the isomer -S and micronized, will present greater bioavailability than hesperidin formed by a mixture of the isomers -S and -R. In turn, the bioavailability of the hesperidin formed mainly by the isomer -S and micronized will present greater bioavailability than the mixture of the isomers -S and -R and micronized.

The main objective of this study was to quantify the bioavailability of three extracts of hesperidin:

* Hesperidin extract with a mixture of the isomers -S and -R.
* Hesperidin extract with a mixture of the isomers -S and -R micronized.
* Hesperidin extract with the isomer -S micronized.

DETAILED DESCRIPTION:
It will be conducted a post-prandial, randomized, crossover, and double-blind nutritional intervention study.

In a first phase, it will be done a pre-selection process with 30 male and female volunteers over 18 years of age. It will be determined hesperidin excreted levels in urine after the consumption of 500 mL of a homogeneous orange juice among all the participants. Sixteen participants will be selected preferably with an intermediate capacity of hesperidin absorption. The aim of this first phase is to obtain a lower variability in the results in the second phase of the study. Of the sixteen participants, six participants will start the study with the consumption of a hesperidin extract, five with the consumption of the second hesperidin extract and five with the consumption of the third hesperidin extract for, after one week washing period, exchange the hesperidin extracts between the three study groups, and finally repeat the exchange of hesperidin extracts after another week of washing period so that, in the total of the study, each participant had consumed the three hesperidin extracts.

Participants will consume two capsules with 250 mg of extract each, being the total orange extract consumed 500 mg, with 450 mg of hesperidin (90%) and the rest (10%) substances coming from the orange in the process of extracting hesperidin.

During the study there will be 5 visits, one selection (V0), one pre-inclusion (V-1) and 3 study visits (V1, V2 and V3).

ELIGIBILITY:
Inclusion Criteria:

1. Men and women over 18 years of age.
2. Firm the informed consent.

Exclusion Criteria:

1. Take supplements or multivitamin supplements or phytotherapeutic products that interfere with the treatment under study up to 30 days before the start of the study.
2. Present intolerances and / or food allergies related to hesperidin.
3. Take antibiotics up to 30 days before the start of the study.
4. Being pregnant or intending to become pregnant.
5. Be in breastfeeding period.
6. Be a smoker
7. Participate in or have participate in a clinical trial or nutritional intervention study in the last 30 days prior to inclusion in the study.
8. Be vegetarian.
9. Present some chronic gastrointestinal disease.
10. Present some chronic disease in clinical manifestation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-06-13 (Actual); Primary Completion 2020-03-02 (Actual); Study Completion 2020-03-02 (Actual)

PRIMARY OUTCOMES:
Bioavailability of hesperidin calculated by urine hesperidin concentration | At week 2, week 3 and week 4.
  Fasting hesperidin metabolites levels in urine will be determined before consuming the capsule with orange extract and in four fractions of time (0-3 hours; 3-6 hours; 6-9 hors and 9-24 hours) until 24 hours postprandially after consuming the capsule.
  The hesperidin levels in urine will be quantified with a Liquid Chromatography (LC)- Mass Spectrometry (MS) equipment.

SECONDARY OUTCOMES:
Area Under The Curve (AUC) of plasma hesperidin levels. | At week 2, week 3 and week 4.
  Fasting hesperidin metabolites levels in blood will be determined before consuming the capsule with orange extract until 24 hours postprandially at 8 points after consuming the capsule (2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 7 hours, 8 hours and 24 hours).
  The hesperidin levels in urine will be quantified with a Liquid Chromatography (LC)- Mass Spectrometry (MS) equipment.
Maximum plasma concentration (Cmax). | At week 2, week 3 and week 4.
  Maximum plasma concentration of hesperidin.
Time for maximum plasma concentration (Tmax). | At week 2, week 3 and week 4.
  Time period for the maximum plasma concentration of hesperidin.
Half-life (T1/2). | At week 2, week 3 and week 4.
  Time taken for half the initial dose of hesperidin administered to be eliminated from the body
Hesperidin catabolites levels in plasma. | At week 2, week 3 and week 4.
  Fasting hesperidin catabolites levels in blood will be determined before consuming the capsule with orange extract until 24 hours postprandially at 8 points after consuming the capsule (2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 7 hours, 8 hours and 24 hours).
  The hesperidin levels in urine will be quantified with a Liquid Chromatography (LC)- Mass Spectrometry (MS) equipment.
Hesperidin catabolites in urine. | At week 2, week 3 and week 4.
  Fasting hesperidin catabolites levels in urine will be determined before consuming the capsule with orange extract and in four fractions of time (0-3 hours; 3-6 hours; 6-9 hors and 9-24 hours) until 24 hours postprandially after consuming the capsule.
  The hesperidin levels in urine will be quantified with a Liquid Chromatography (LC)- Mass Spectrometry (MS) equipment.
Quantification of hesperidin bioavailability for the selection of individuals | At week 1.
  For the selection of intermediate hesperidin absorption individuals fasting hesperidin metabolites levels in urine will be determined before consuming 500 ml of an orange juice and in 24 hours postprandially after consuming the orange juice.
  The hesperidin levels in urine will be quantified with a Liquid Chromatography (LC)- Mass Spectrometry (MS) equipment.

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Solà, Dr, Principal Investigator — Centro Tecnológico de Nutrición y Salud (Eurecat_Reus). Reus, Tarragona, Spain.
Locations (1):
- Centro Tecnológico de Nutrición y Salud (Eurecat-Reus), Reus, Tarragona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Technological Centre of Nutrition and Health. Eurecat_Reus. — http://eurecat.org